CLINICAL TRIAL: NCT00677638
Title: Catheter-Based Transapical Implantation of the Ventor Embracer™ Heart Valve Prosthesis in Patients With Severe Aortic Valve Disease
Brief Title: Transapical Implantation of Ventor Embracer™ Valve in Patients With Severe Aortic Valve Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Ventor Technologies (Industry)
Responsible Party: Sharon Sax, Ventor Technologies
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLIN004
Record Dates: First submitted 2008-05-12; First posted 2008-05-14 (Estimated); Last update posted 2009-12-03 (Estimated); Status verified 2009-12

CONDITIONS: Aortic Valve Disease
MeSH Terms: conditions — Aortic Valve Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Embracer implantation
  Interventions: Device: Ventor Embracer

INTERVENTIONS:
Device: Ventor Embracer — Implantation of Ventor Embracer

SUMMARY:
A prospective single arm study evaluating feasibility and safety of a catheter-based transapical implantation of the Ventor Embracer™ aortic valve bioprosthesis in patients with severe aortic valve disease, specifically aortic stenosis, who are at elevated risk for standard surgical valve replacement.

ELIGIBILITY:
Inclusion Criteria:

1. Patient understands the implications of participating in the study and provides informed consent
2. Patient is willing to comply with specified follow-up evaluation and can be contacted by telephone
3. Age >75 years
4. Severe, aortic stenosis (echocardiographically derived mean gradient > 40 mm Hg, and/or jet velocity > 4m/s, or an initial aortic valve area of < 0.8 cm2)
5. Symptoms related to the aortic valve disease, as demonstrated by NYHA Functional Class II or greater
6. EuroSCORE scale of >9 points indicating a predicted risk for mortality of >11% according to the logistic EuroSCORE
7. Echocardiographically determined anteroposterior aortic annulus diameter of >19 and <23 mm
8. Echocardiographically determined sinotubular junction diameter of ≥23 mm

Exclusion Criteria:

1. Congenital unicuspid or bicuspid aortic valve
2. Fused commissures
3. Severe eccentricity of calcification
4. Echocardiographic evidence of intracardiac mass, thrombus, or vegetation.
5. Severe left ventricular dysfunction (LVEF < 25%)
6. More than mild right ventricular dysfunction
7. Hypertrophic obstructive cardiomyopathy
8. Moribund patients, or patients with a noncardiac disease limiting by itself life expectancy to less than 12 months
9. Known hypersensitivity or contraindication to any study medication
10. Known sensitivity to contrast medium that cannot be adequately controlled with pre-medication
11. Known allergy or sensitivity to Nitinol
12. Sepsis, or acute endocarditis
13. Blood dyscrasia such as acute anemia, leucopenia, or thrombocytopenia; bleeding diathesis, or coagulopathy.
14. Renal insufficiency and/or end stage renal disease requiring chronic dialysis
15. Liver disease as indicated by jaundice, ascites, ALT/AST > 3 x ULN, elevation of total bilirubin > 1.5 mg/dl, albumin < 3.0 g/l, or INR > 1.5 (if not on anticoagulation).
16. Significant lung disease (e.g. FEV1 < 1.2L or FEV1 < 50%).
17. Active peptic ulcer or GI bleeding within 3 months from the planned index procedure
18. Untreated clinically significant coronary artery disease requiring revascularisation
19. Cardiogenic shock, suspected cardiogenic shock, or hemodynamic instability requiring inotropic support or mechanical heart assistance
20. Peripheral vascular disease, including abdominal and thoracic aortic disease, which could pose a problem for eventual transarterial mechanical support (e.g. Intraaortic Balloon Pump)
21. Need for emergency surgery, cardiac or noncardiac
22. History of myocardial infarction in the last 6 weeks.
23. History of TIA or stroke in the last 6 months.
24. Any therapeutic invasive cardiac procedure, except aortic balloon valvuloplasty, performed within 30 days from the planned index procedure, or 6 months, in case of implantation of drug-eluting stents.
25. Uncontrolled atrial fibrillation
26. Pre-existing aortic valve replacement
27. Severe (greater than 3+) mitral regurgitation
28. Severe (greater than 3+) aortic regurgitation
29. Patient is currently enrolled in another investigational device or drug trial

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2008-06; Primary Completion 2010-01 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Stable device placement and adequate function as assessed by angiography and echocardiography immediately post-procedure | day one
A composite of any death, myocardial infarction, or disabling stroke at 30 days post-procedure | 30 days

SECONDARY OUTCOMES:
Device success and the absence of periprocedural MACCEs at post-operative day 1 | day one
Any of the following adverse events: death, myocardial infarction, disabling stroke, repeat aortic valve procedure, cardiogenic shock, or endocarditis at 30 days | 30 days
Any of the following adverse events: death, disabling stroke, repeat aortic valve procedure or endocarditis at 6 months | 6 months
Freedom from death at 1 year | 1 year
Functional improvement from baseline per New York Heart Association (NYHA) functional classification at 30 days, 6 months and 1 year | 1 year
Peak & mean pressure gradient, derived calculated measures of prosthetic valve function, aortic regurgitation - assessed by echocardiography immediately after deployment, at POD 1, 30 days, 6 months and 5 years annually | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Jochen Schaefers, MD, Principal Investigator — Universitatsklinikum des Saarlandes; Friedrich Mohr, MD, Principal Investigator — Universität Leipzig
Locations (3):
- Germany (3):
  - Prof. Thorsten Wahlers, Cologne
  - Prof. Jochen Schaefers, Homburg
  - Friedrich Mohr, MD, Leipzig

REFERENCES:
- [Derived] Falk V, Walther T, Schwammenthal E, Strauch J, Aicher D, Wahlers T, Schafers J, Linke A, Mohr FW. Transapical aortic valve implantation with a self-expanding anatomically oriented valve. Eur Heart J. 2011 Apr;32(7):878-87. doi: 10.1093/eurheartj/ehq445. Epub 2010 Dec 9. PMID 21148541